CLINICAL TRIAL: NCT07218185
Title: Comparative Effectiveness of Pathogen Reduced Cryoprecipitated Fibrinogen Complex (INTERCEPT Fibrinogen Complex, IFC) and Cryoprecipitate-AHF (Cryo-AHF) for Treatment of Trauma Associated Hemorrhage: CRYO-FIRST, A Quality Improvement Study
Brief Title: Comparative Effectiveness of INTERCEPT Fibrinogen Complex (IFC) and Cryoprecipitate-AHF (Cryo-AHF) for Treatment of Trauma Associated Hemorrhage
Acronym: CRYO-FIRST
Status: Not yet recruiting | Type: Observational
Sponsor: Cerus Corporation (Industry)
Collaborators: Coalition for National Trauma Research (Other)
Responsible Party: Sponsor
Other Study IDs: CLI 00193
Record Dates: First submitted 2025-09-30; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hypofibrinogenemia; Hemorrhage
Keywords: Fibrinogen; Hemorrhage; Trauma; Resuscitation
MeSH Terms: conditions — Afibrinogenemia; Hemorrhage; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IFC arm: Subjects will receive Pathogen Reduced Cryoprecipitated Fibrinogen Complex (IFC) for fibrinogen supplementation.
  Interventions: Biological: Pathogen Reduced Cryoprecipitated Fibrinogen Complex
- Cryo AHF arm: Subjects will receive Cryoprecipitated-Antihemophilic Factor (Cryo-AHF) for fibrinogen supplementation.
  Interventions: Biological: Cryoprecipitated-Antihemophilic Factor

INTERVENTIONS:
Biological: Pathogen Reduced Cryoprecipitated Fibrinogen Complex — IFC will be administered based on the study site's assigned treatment block. Study subjects will receive IFC with a point-of-care testing value of FCS <1.6 hPa. Additional IFC may be administered per point-of-care testing or clinical judgement, as needed.
  Other Names: INTERCEPT Fibrinogen Complex; IFC
  Groups: IFC arm
Biological: Cryoprecipitated-Antihemophilic Factor — Cryo-AHF will be administered based on the study site's assigned treatment block. Study subjects will receive Cryo-AHF with a point-of-care testing value of FCS <1.6 hPa. Additional Cryo-AHF may be administered per point-of-care testing or clinical judgement, as needed.
  Other Names: Cryo-AHF; Cryoprecipitate-AHF; Cryo
  Groups: Cryo AHF arm

SUMMARY:
The objective of this study is to determine the feasibility and effectiveness of early IFC administration in patients with functional hypofibrinogenemia associated with hemorrhagic shock (HS). This study will elucidate whether advancements in rapid testing for functional hypofibrinogenemia and provision of a shelf-stable fibrinogen complex (IFC) results in a shorter time to administration of fibrinogen replacement, thus overcoming the limitations encountered by prior trials.

This study aims to:

* Demonstrate the feasibility and response to early administration of pre-thawed IFC compared to CRYO-AHF when ordered during resuscitation of severely injured patients with HS and functional hypofibrinogenemia.
* Assess effectiveness of early administration of pre-thawed IFC vs CRYO-AHF in severely injured patients with HS and functional hypofibrinogenemia on proximate process measures of resuscitation.
* Assess clinical outcomes in severely injured patients with HS and functional hypofibrinogenemia receiving early administration of pre-thawed IFC vs CRYO-AHF product.

DETAILED DESCRIPTION:
This study is a multicenter, multi-period, by hospital cluster randomized, alternating treatment block crossover study comparing pre-thawed Pathogen Reduced Cryoprecipitated Fibrinogen Complex (INTERCEPT Fibrinogen Complex, IFC) to Cryoprecipitate-AHF (Cryo-AHF) in patients with hemorrhagic shock and functional hypofibrinogenemia.

This study will assess the feasibility and effectiveness of early IFC administration in trauma patients in hemorrhagic shock with functional hypofibrinogenemia. Specifically, it aims to determine whether IFC enables faster delivery of fibrinogen replacement compared to Cryo-AHF and equivalent correction of hypofibrinogenemia. Currently, the use of IFC vs Cryo-AHF varies by center and blood bank availability, and both are considered standard-of-care treatment options. This study evaluates their performance in routine clinical use.

The primary outcomes are the proportion of patients who receive fibrinogen replacement within 60 minutes of arrival; and the correction of functional hypofibrinogenemia. Secondary outcomes include proximate measures of resuscitation including time to hemostasis, estimated blood loss, blood transfusion burden, 3-hour, 6-hour, 24-hour and 30-day mortality and adverse event incidences including: adult respiratory distress syndrome, multiple organ dysfunction, venous thromboemboli, acute kidney injury, sepsis and transfusion related acute lung injury.

Patients ≥18 years old, or >50 Kg if age unknown, arriving within one hour of estimated time of injury with signs of hemorrhagic shock, will be screened and arrival hypofibrinogenemia determined using the point-of care Quantra® Hemostasis Analyzer. Eligible patients will receive either IFC or Cryo-AHF, depending on site assignment, in alternating 6-month treatment clusters. A post-treatment assessment of fibrinogen will be performed to assess response to fibrinogen supplementation. All data will be collected through 30 days, discharge, or death, whichever occurs first. Four Level 1 trauma centers will enroll a total of 320 patients (estimated each center to enroll approximately 80 patients) over 24 months of the study. If a site under-recruits, other sites may increase recruitment with IRB approval.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic injury
* Age ≥18 years or estimated weight ≥ 50 kg, if age unknown
* Presenting to participating trauma center ≤1 hour from estimated time of injury
* Functional hypofibrinogenemia upon arrival to the trauma center as measured by POC testing (Quantra) with an FCS < 1.6 hPa
* Hemorrhagic shock defined as:

  1. Initiation of transfusion of any uncross matched blood product AND
  2. Evidence of active hemorrhage as judged by the attending trauma surgeon AND
  3. Initiation of the participating trauma center's MTP
* IFC or CRYO-AHF are available at the time of enrollment.

Exclusion Criteria:

* Suspected isolated severe brain or spinal cord injury
* Isolated drowning or hanging
* Burns > 20% total body surface area (TBSA)
* Known pregnancy
* Admitted from a correctional facility
* Known do not resuscitate (DNR) order
* Traumatic arrest >5 minutes
* Isolated fall from standing
* Emergency Department (ED) thoracotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemorrhagic trauma
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Correction of functional fibrinogen | From time of initiation of anesthesia until time of completion of resuscitation.
  The correction of functional fibrinogen as measured by point-of-care testing (Quantra) after transfusion of IFC or CRYO-AHF, as measured at completion of resuscitation. The time to correction of functional fibrinogen is reported in hours and minutes.
The proportion (%) of patients who receive IFC or Cryo-AHF within 60 minutes of presentation to the participating trauma center. | From time of admission to the hospital trauma service to initial transfusion of either IFC or Cryo-AHF, measured in hours and minutes.
  The proportion (%) of patients with hemorrhagic shock who have functional hypofibrinogenemia and who receive IFC or Cryo-AHF within 60 minutes of presentation to the participating trauma center.

SECONDARY OUTCOMES:
Mortality rates | Measured from the time of admission to the hospital trauma service until death. Measured at 3, 6, and 24 hours after admission and reported in hours. Beyond 24 hours and up to 30 days post-admission, mortality is measured and reported in days.
  Mortality rates at 3, 6, 24 hours and 30 days.
Clinical complications | Within 24 hours of treatment.
  Incidences of adverse events to include Acute blood loss anemia, Abdominal compartment syndrome, Acute Kidney Injury, Acute Renal Failure, Acute respiratory distress syndrome, Bleeding after hemostasis requires intervention, Coagulopathy, Febrile non-hemolytic transfusion reaction, Hospital Acquired Pneumonia, Intraabdominal infection, Liver Failure, multiple organ dysfunction (MOD), Multiple Organ Failure (MOF), Myocardial infarction, Sepsis, Stroke, Surgical Site infection, Symptomatic and asymptomatic deep vein thrombosis, Symptomatic and asymptomatic pulmonary embolism, Systemic Inflammatory Response Syndrome, Transfusion-associated circulatory overload (TACO), Transfusion-associated lung injury (TRALI), Transfusion-related allergic reactions, Transfusion-related hyperkalemia (in first 24hrs), Transfusion-related hypocalcemia (in first 24hrs, and Ventilator-associated pneumonia.

OTHER OUTCOMES:
Time to hemostasis (TTH) | From time of admission to the trauma service until either hospital day 30, day of discharge, or death, whichever comes first, for a maximum of 30 days.
  Measurement of the time until cessation of bleeding. Cessation of bleeding is determined by the surgeon by visual inspection or the patient requiring no transfusion for ≥1 hour.
Time to Completion of Resuscitation (COR) | From time of initiation of the MTP by the trauma service (measured in hours and minutes) until discontinuation of the MTP until either hospital day 30, day of discharge or death, whichever comes first, for a maximum of 30 days.
  Measurement of the time (reported in hours and minutes) of COR as determined by the discontinuation of the massive transfusion protocol (MTP) and achievement of anatomic hemostasis (no further bleeding from injured blood vessels and organs with adequate blood flow) determined by visual inspection.
Total volume of resuscitation (TVOR) | From time of admission to the hospital trauma service, measured at 24 hours after admission, and measured at COR at either hospital day 30, day of discharge, or death, whichever comes first, for a maximum of 30 days.
  Measurement of the total volume (measured in mL) of blood products administered within the first 24 hours after admission to the hospital trauma service and until time of complete resuscitation (COR) as determined by the discontinuation of the massive transfusion protocol (MTP) and cessation of bleeding from damaged blood vessels and organs with adequate blood flow.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado, Anschutz Medical Center, Aurora, Colorado
  - Jackson Memorial Hospital, University of Miami, Miami, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Barnes-Jewish Hospital, Washington University of Saint Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.nattrauma.org

REFERENCES:
- [Result] Rossetto A, Wohlgemut JM, Brohi K, Davenport R. Sonorheometry versus rotational thromboelastometry in trauma: a comparison of diagnostic and prognostic performance. J Thromb Haemost. 2023 Aug;21(8):2114-2125. doi: 10.1016/j.jtha.2023.04.031. Epub 2023 May 8. PMID 37164268
- [Result] Huffman G, Wilken N, Loh JH, Fazal M, Lei I, Myers A, et al. Analysis of Wastage, Savings, and Maternal and Pediatric Outcomes for Pooled Pathogen Reduced Cryoprecipitate versus Conventional Cryoprecipitate. Baylor College of Medicine; Abstract AABB Annual Meeting. 2024.
- [Result] Holcomb JB, Tilley BC, Baraniuk S, Fox EE, Wade CE, Podbielski JM, del Junco DJ, Brasel KJ, Bulger EM, Callcut RA, Cohen MJ, Cotton BA, Fabian TC, Inaba K, Kerby JD, Muskat P, O'Keeffe T, Rizoli S, Robinson BR, Scalea TM, Schreiber MA, Stein DM, Weinberg JA, Callum JL, Hess JR, Matijevic N, Miller CN, Pittet JF, Hoyt DB, Pearson GD, Leroux B, van Belle G; PROPPR Study Group. Transfusion of plasma, platelets, and red blood cells in a 1:1:1 vs a 1:1:2 ratio and mortality in patients with severe trauma: the PROPPR randomized clinical trial. JAMA. 2015 Feb 3;313(5):471-82. doi: 10.1001/jama.2015.12. PMID 25647203
- [Result] Davenport R, Curry N, Fox EE, Thomas H, Lucas J, Evans A, Shanmugaranjan S, Sharma R, Deary A, Edwards A, Green L, Wade CE, Benger JR, Cotton BA, Stanworth SJ, Brohi K; CRYOSTAT-2 Principal Investigators. Early and Empirical High-Dose Cryoprecipitate for Hemorrhage After Traumatic Injury: The CRYOSTAT-2 Randomized Clinical Trial. JAMA. 2023 Nov 21;330(19):1882-1891. doi: 10.1001/jama.2023.21019. PMID 37824155
- [Result] Curry N, Rourke C, Davenport R, Beer S, Pankhurst L, Deary A, Thomas H, Llewelyn C, Green L, Doughty H, Nordmann G, Brohi K, Stanworth S. Early cryoprecipitate for major haemorrhage in trauma: a randomised controlled feasibility trial. Br J Anaesth. 2015 Jul;115(1):76-83. doi: 10.1093/bja/aev134. Epub 2015 May 19. PMID 25991760
- [Result] McQuilten ZK, Bailey M, Cameron PA, Stanworth SJ, Venardos K, Wood EM, Cooper DJ. Fibrinogen concentration and use of fibrinogen supplementation with cryoprecipitate in patients with critical bleeding receiving massive transfusion: a bi-national cohort study. Br J Haematol. 2017 Oct;179(1):131-141. doi: 10.1111/bjh.14804. Epub 2017 Jun 27. PMID 28653339
- [Result] Holcomb JB, del Junco DJ, Fox EE, Wade CE, Cohen MJ, Schreiber MA, Alarcon LH, Bai Y, Brasel KJ, Bulger EM, Cotton BA, Matijevic N, Muskat P, Myers JG, Phelan HA, White CE, Zhang J, Rahbar MH; PROMMTT Study Group. The prospective, observational, multicenter, major trauma transfusion (PROMMTT) study: comparative effectiveness of a time-varying treatment with competing risks. JAMA Surg. 2013 Feb;148(2):127-36. doi: 10.1001/2013.jamasurg.387. PMID 23560283